CLINICAL TRIAL: NCT06805292
Title: Evaluation of Acacia Catechu and Low-Level Laser in the Treatment of Stage II Periodontitis
Brief Title: Evaluation of Acacia Catechu and Low-Level Laser in the Treatmentof Stage II Periodontitis
Acronym: LLLvsAgel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Dental Medicine for Girls (Other Government)
Responsible Party: Principal Investigator, Mona Monsour, Master's degree student at Oral Medicine, Periodontology, Oral Diagnosis, and Oral Radiology Department, Faculty of Dental Medicine for Girls, Al-Azhar University., Principal Investigator)., Faculty of Dental Medicine for Girls
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMPDR-108-1J
Record Dates: First submitted 2024-12-30; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Chronic Periodontitis
Keywords: Chronic periodontitis; Herbal Medicine; Low Level Laser Therapy; Adjunctive therapy; Acacia catechu
MeSH Terms: conditions — Chronic Periodontitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Groupe (Active Comparator): treated with non-surgical periodontal therapy and serves as a control group.
  Interventions: Other: phase 1 therapy chronic periodontitis
- Test: Acacia gel group (Active Comparator): using A. catechu gel adjunctive to non-surgical periodontal therapy
  Interventions: Other: Acacia catechu
- Test: laser group (Active Comparator): Group III: using low-level laser adjunctive to non-surgical periodontal therapy.
  Interventions: Other: Low Level Laser Therapy
- Test: Acacia gel +laser group (Active Comparator): Group IV: using A. catechu gel with low-level laser adjunctive to non-surgical periodontal therapy.
  Interventions: Other: Acacia catechu; Other: Low Level Laser Therapy; Other: phase 1 therapy chronic periodontitis; Other: local drug delivary acacia +LLL

INTERVENTIONS:
Other: Acacia catechu — local delivery of acacia catechu gel in patient with chronic periodontitis stage 2
  Other Names: acaia catech gel; black catechu (trade name ); black cutch; cutch tree,; gel of aqueous extract of A.catechu bark
  Arms: Test: Acacia gel +laser group; Test: Acacia gel group
Other: Low Level Laser Therapy — low-level laser as an adjunctive therapy in patient with chronic periodontitis stage 2
  Other Names: Biomodulation
  Arms: Test: Acacia gel +laser group; Test: laser group
Other: phase 1 therapy chronic periodontitis — patient with chronic periodontitis stage 2 will go for phase one therapy only
  Other Names: phase 1 therapy (scalling +root planning)
  Arms: Control Groupe; Test: Acacia gel +laser group
Other: local drug delivary acacia +LLL — pateient with chronic periodontitis treated with LLL +acacia catehu gel
  Other Names: LLL +acacia catehu gel
  Arms: Test: Acacia gel +laser group

SUMMARY:
Evaluation of Acacia catechu and Low-Level Laser in the Treatment of Stage 2 Periodontitis.

DETAILED DESCRIPTION:
* Assess the effectiveness of A. catechu gel (local delivery) adjunctive to non surgical therapy in the treatment of stage chronic periodontitis. Clinical and biochemical evaluation.
* Compare the effectiveness of A. catechu gel (local delivery) and low-level laser adjunctive to non-surgical therapy in the treatment of stage chronic periodontitis.

Clinical and biochemical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Motivated patient with good oral hygiene.
2. Age ranges from (30-50) years.
3. Free from any systemic disease according to the Cornell Medical Index (16).

Exclusion Criteria:

1. Patients who received periodontal treatment over the 12 months preceding the study.
2. Patients who consumed antibiotics or anti-inflammatory drugs within the last 3 months.
3. Previous or current radiation or immunosuppressive therapies.
4. Pregnant & lactating women.
5. Patient with orthodontic appliances. Or having partial dentures.
6. Patient with parafunctional habits.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
inflammatory biomarker | 0 and 6 month evaluation
  Measuring Interleukin 1 beta level
Antioxidant biomarker | 0 and 6 month evaluation
  measuring total antioxidant capacity.

SECONDARY OUTCOMES:
gingival index | 0,1,3,6 month evaluation
  clinical evaluation of GI
  score from (0 to 3) 0 = normal is the best value. 3 = diseesed (the worst value).
  0=Normal gingiva.
  1. = mild inflammation, a slight change in color, slight edema, no bleeding on probing.
  2. = moderate inflammation, redness, edema, and glazing; bleeding on probing.
  3. = severe inflammation, marked redness and edema, ulceration, and the tendency to spontaneous bleeding.
clinical attachment level or loss | 0,1,3,6 month evaluation
  * Clinical Attachment Level (CAL) or loss: Clinical attachment level was measured from the cementoenamel junction to the base of the pocket using a University of Michigan probe with the University of North Carolina periodontal probe (UNC15) around each tooth.
  * measurement unite by millimetre
  * zero clinical attachment level means no periodontitis
  * clinical attachment loss is a critical parameter differentiated betwwn gingivitis and periodontitis
  * the less the number, the better the case improvement.
  * cal of 2 mm is better than cal of 4 mm.
plaque index | 0,1,3,6 month evaluation
  evaluation of PI score from (0-3) 0 is the best value; 3 is the worst.
  0=No plaque is visible, even when a probe is used.
  1. = Some plaque is visible only when a probe is used to skim the tooth surface.
  2. = A visible amount of plaque can be seen without a probe.
  3. = abudant amount of plaque at gingival margin, interdental spaces filled with plaque.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Gawish, professor, Study Director — Al-Azhar University; mostafa hegazy, professor, Study Director — Al-Azhar University
Locations (1):
- Mona Mansour, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No